CLINICAL TRIAL: NCT04762420
Title: Sugammadex Dosing: Anaesthesiologist Clinical Perception Versus Quantitative Monitoring
Status: Completed | Type: Observational
Sponsor: Hospital do Divino Espírito Santo de Ponta Delgada (Other)
Responsible Party: Principal Investigator, Ernesto Ruivo, Principal Investigator, Hospital do Divino Espírito Santo de Ponta Delgada
Other Study IDs: DivinoEspíritoSanto
Record Dates: First submitted 2021-02-10; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Neuromuscular Blockade; Anesthesia; TOF; Curarization, Postoperative Residual
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sugammadex dose as suggested by senior anaesthesiologists (SSD) based on clinical experience.
  Interventions: Other: Dose of sugammadex according to SSD and QSD
- Dose of Sugammadex determined by quantitative monitoring (QSD).
  Interventions: Other: Dose of sugammadex according to SSD and QSD

INTERVENTIONS:
Other: Dose of sugammadex according to SSD and QSD — At the time of pharmacologic reversal of the NMB, both the SSD and QSD, according to portuguese guidelines on the management of the NMB, were recorded. The QSD was then administered to the patient. The SSD was considered appropriate if it was within 10% of the recommended dose for the given depth of NMB, as measured by TOFscan® monitor. The results were analyzed descriptively.

SUMMARY:
Many clinicians continue to rely on subjective evaluation in making decisions about the adequacy of neuromuscular function before tracheal extubation rather than using quantitative monitoring. The aim was to compare the sugammadex dose as suggested by senior anaesthesiologists (SSD) based on clinical experience versus the dose determined by quantitative monitoring (QSD) to determine if the subjective dose was appropriate.

DETAILED DESCRIPTION:
Materials and Methods:

After obtaining approval from the Institute Ethics Committee, a prospective 3-month study in patients aged 18-75 years who underwent general anesthesia with rocuronium (initial dose 0.6 mg/kg) NMB and subsequent reversal with sugammadex, was carried out. American Society of Anesthesiologists (ASA ) physical status V, emergency surgery, patients with hypersensitivity history to rocuronium or sugammadex, severe renal impairment/dialysis, neuromuscular diseases, severe hepatic disease, pre-existing coagulopathies and pregnancy were excluded. Monitoring included ASA standard monitoring, bispectral index and NMB monitoring using TOFscan® monitor. The senior anaesthesiologist was blinded to the TOFscan®, which was only available to the author.

At the time of pharmacologic reversal of NMB, both the sugammadex dose proposed by the anaesthesiologist (SSD) and the dose suggested by TOFscan® (QSD) according to the Portuguese recommendations for the management of NMB were recorded. Afterwards the QSD was administered to overcome ethical issues. When train-of-four (TOF) count was 0, the author performed the post tetanic count (PTC) stimulus to determine the recommended dose. The SSD was considered appropriate if it was within 10% of the QSD for the depth of NMB. All patients were extubated with a TOF ratio > 0.9 (TOFr) and both the rocuronium and sugammadex dose were calculated based on the real patient weight. Data regarding anaesthesia, duration of anaesthesia and dosing pattern of rocuronium were also noted. The results were analysed descriptively.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years;
* Above patients who underwent general anesthesia with rocuronium neuromuscular blockade and subsequent reversal with sugammadex.

Exclusion Criteria:

* American Society of Anesthesiologists physical status V;
* Emergency surgery;
* Hypersensitivity history to rocuronium or sugammadex;
* Severe renal impairment/dialysis;
* Neuromuscular diseases;
* Severe hepatic disease;
* Pre-existing coagulopathies;
* Pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population was made of 66 individuals, aged 18-75 years who underwent general anesthesia with rocuronium (initial dose 0.6 mg/kg) neuromuscular blockade and subsequent reversal with sugammadex.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
The percentage of patients who would receive an adequate or inadequate (over or under) dose of sugammadex. | 3 months
  Given the interindividual variability response to neuromuscular block, which makes it difficult to subjectively determine the dose needed, the aim was to compare the sugammadex dose as suggested by senior anaesthesiologists based on clinical experience versus the dose determined by quantitative monitoring to determine if the subjective dose was appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Frias, MD, Principal Investigator — Hospital do Divino Espírito Santo de Ponta Delgada
Locations (1):
- Hospital do Divino Espírito Santo, Ponta Delgada, Portugal

IPD SHARING:
Plan to Share IPD: No
Prospective, 3-month study in 66 patients aged 18-75 years who underwent general anesthesia with rocuronium neuromuscular block and reversal with sugammadex.

REFERENCES:
- [Result] Esteves S, Roxo A, Resendes H, Pereira L, Fernandes N, Borges S. Recomendações Portuguesas para a Gestão do Bloqueio Neuromuscular 2017. Rev Soc Port Anestesiol. 2018; 27: 4-52.
- [Result] Dutu M, Ivascu R, Tudorache O, Morlova D, Stanca A, Negoita S, Corneci D. Neuromuscular monitoring: an update. Rom J Anaesth Intensive Care. 2018 Apr;25(1):55-60. doi: 10.21454/rjaic.7518.251.nrm. PMID 29756064
- [Result] Unterbuchner C. Neuromuscular Block and Blocking Agents in 2018. Turk J Anaesthesiol Reanim. 2018 Apr;46(2):75-80. doi: 10.5152/TJAR.2018.200318. Epub 2018 Apr 1. No abstract available. PMID 29744239
- [Result] Naguib M, Brull SJ, Johnson KB. Conceptual and technical insights into the basis of neuromuscular monitoring. Anaesthesia. 2017 Jan;72 Suppl 1:16-37. doi: 10.1111/anae.13738. PMID 28044330
- [Result] Cammu G. Sugammadex: Appropriate Use in the Context of Budgetary Constraints. Curr Anesthesiol Rep. 2018;8(2):178-185. doi: 10.1007/s40140-018-0265-6. Epub 2018 Mar 20. PMID 29904285
- [Result] Ciara Mitchell, Steve Lobaz. An Overview of Sugammadex. ATOTW 332 (2016); 1-6
- [Result] Daniel Moi. Residual Neuromuscular Blockade, ATOTW 290 (2013); 1-8
- [Result] A. Castagnoli, M. Adversi, G. Innocenti, G.F. Di Nino and R.M. Melotti. Post-Operative Residual Curarization (PORC): A Big Issue for Patients' Safety. Risk Management for the Future - Theory and Cases, 2012, 117-136
- [Result] Wycherley AS, Bembridge JL. Monitoring techniques; neuromuscular blockade and depth of anaesthesia. Anaesthesia and intensive care medicine (2017).
- [Result] Syed F, Trifa M, Uffman JC, Tumin D, Tobias JD. Monitoring of Sugammadex Dosing at a Large Tertiary Care Pediatric Hospital. Pediatr Qual Saf. 2018 Oct 9;3(5):e113. doi: 10.1097/pq9.0000000000000113. eCollection 2018 Sep-Oct. PMID 30584640
- [Result] Takazawa T, Katsuyuki M, Sawa T, et al. The current status of sugammadex usage and the occurrence of sugammadex-induced anaphylaxis in Japan. APSF Newsletter 2018;33:1.
- [Result] Goltz K, Dambach M, Schlapfer M, Biro P. Non-Feasibility to Estimate the Need for Reversal of Neuromuscular Relaxation from the Applied Rocuronium Dosing Pattern: A Retrospective Analysis of Anaesthesia Records. Turk J Anaesthesiol Reanim. 2018 Feb;46(1):57-61. doi: 10.5152/TJAR.2018.98705. Epub 2018 Feb 1. PMID 30140502
- [Result] de Boer HD, Carlos RV, Brull SJ. Is lower-dose sugammadex a cost-saving strategy for reversal of deep neuromuscular block? Facts and fiction. BMC Anesthesiol. 2018 Nov 6;18(1):159. doi: 10.1186/s12871-018-0605-6. PMID 30400850